CLINICAL TRIAL: NCT06727565
Title: VELOCITY-HNSCC Substudy-01: A Phase 2 Study of Novel Combination Therapies in Participants With Previously Untreated Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma Regardless of PD-L1 Expression Status
Brief Title: Study of Novel Treatment Combination Therapies in Participants With Head and Neck Squamous Cell Carcinoma Regardless of PD-L1 Expression Status; Substudy-01
Acronym: VELOCITY-HNSCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Arcus Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-699-7184-01; 2024-513121-22 (Other: EU Trial (CTIS) Number)
Record Dates: First submitted 2024-12-09; First posted 2024-12-11 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — zimberelimab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Group A: Domvanalimab (DOM) + Zimberelimab (ZIM) + Platinum-based Chemotherapy (Experimental): Participants will receive DOM + ZIM + platinum-based chemotherapy (paclitaxel + carboplatin).
  Interventions: Drug: Domvanalimab; Drug: Zimberelimab; Drug: Paclitaxel; Drug: Carboplatin
- Treatment Group B: Zimberelimab (ZIM) + Platinum-based Chemotherapy (Experimental): Participants will receive ZIM + platinum-based chemotherapy (paclitaxel + carboplatin).
  Interventions: Drug: Zimberelimab; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Domvanalimab — Administered intravenously
  Arms: Treatment Group A: Domvanalimab (DOM) + Zimberelimab (ZIM) + Platinum-based Chemotherapy
Drug: Zimberelimab — Administered intravenously
Drug: Paclitaxel — Administered intravenously
Drug: Carboplatin — Administered intravenously

SUMMARY:
Master protocol: The main goal of this master clinical study is to evaluate the efficacy and safety of multiple novel combination therapies in participants with head and neck squamous cell carcinoma (HNSCC) in various substudies.

Substudy-01 will evaluate the efficacy and safety of novel combination of treatment regimens, domvanalimab (DOM) and zimberelimab (ZIM) combined with chemotherapy vs ZIM combined with chemotherapy.

The primary objective is to assess the efficacy of DOM and ZIM in combination with chemotherapy versus ZIM in combination with chemotherapy.

DETAILED DESCRIPTION:
This platform study will begin with a substudy targeting first-line (1L) recurrent or metastatic (r/m) HNSCC regardless of programmed cell death ligand 1 (PD-L1) expression status (Substudy-01), and new substudies may be added in the future targeting different study populations of HNSCC. All substudies evaluating additional drugs will be added in a staggered manner when relevant nonclinical and/or clinical data become available. Additional drugs may also be added to Substudy-01 in the future.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically or cytologically confirmed r/m squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, and larynx that is considered incurable by local therapies.
* No prior systemic therapy for r/m HNSCC. Individuals who had disease progression or recurrence more than 6 months after the last dose of curative intent systemic platinum-containing therapy for locoregionally advanced disease are eligible.
* At least 1 measurable lesion by computed tomography or magnetic resonance imaging that qualifies as a RECIST v1.1 target lesion at baseline.
* Have adequate tumor tissue samples preferably from lesions not irradiated prior to biopsy (acceptable from irradiated lesions if disease progression has been demonstrated in such lesions) to submit for central testing.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Known results from human papillomavirus (HPV) status test (p16 expression) for oropharyngeal carcinoma defined as p16 testing.

Key Exclusion Criteria:

* Individuals with nasopharyngeal cancer (any histology), squamous cell carcinoma of unknown primary tumors, skin (cutaneous squamous cell carcinoma), paranasal sinuses, and salivary gland.
* Have disease that is suitable for any local therapies with curative intent.
* Individuals who had disease progression or recurrence within 6 months after the last dose of curative intent systemic platinum-containing therapy for locoregionally advanced disease.
* Have a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Have an active autoimmune disease that required systemic treatment in the past 2 years. (ie, with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
* Prior treatment with any of the following within the specific time frame prior to the first dose of study drug:

  * Major surgery for any cause or significant traumatic injury within 4 weeks prior to the first dose of study drug. Individuals must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study drug.
  * Any noninvestigational anticancer therapy (chemotherapy, biologic therapy, targeted therapy, hormone therapy, or immunotherapy, etc) within 4 weeks prior to the first dose of study drug. Concurrent use for noncancer related condition (eg, hormone replacement therapy) is acceptable.
  * Any investigational drugs (drugs not marketed for any indication) within 4 weeks or 5 half-lives (whichever is longer) prior to the first dose of study drug.
  * Radiation therapy within 2 weeks prior to the first dose of study drug. Individuals must have recovered to Grade ≤ 1 from all radiation-related toxicities, not requiring corticosteroid, and have not experienced radiation pneumonitis.
* Received prior treatment with any anti-PD-1/PD-L1, anti-TIGIT, or other immune checkpoint inhibitors.
* Currently receiving chronic systemic steroids (> 10 mg/day prednisone or its equivalent). Use of topical, inhalational, intranasal, intraocular steroids, and use as premedication for hypersensitivity reactions (eg, IV contrast allergy) are permitted.
* Any unresolved toxicity (Grade ≥ 2) per National Cancer Institute Common Terminology Criteria for Adverse Events v5.0 from prior anticancer therapy or surgical intervention, with the exception of alopecia, vitiligo, and the laboratory toxicities if the laboratory thresholds defined in the inclusion criteria are met. Individuals with Grade ≤ 2 neuropathy are eligible for this study.
* Have an active second malignancy or have had an active second malignancy within 3 years prior to enrollment.
* Have known active central nervous system (CNS) metastases. Individuals with previously treated brain metastases may participate provided they have stable CNS disease for at least 4 weeks prior to enrollment and all neurologic symptoms have returned to baseline, have no evidence of new or enlarging brain metastasis and are not requiring use of steroid for at least 14 days prior to the first dose of study drugs.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 36 months
  ORR is defined as the proportion of participants who achieve a complete response (CR) or partial response (PR) as measured by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 using investigator assessments.
Progression-free survival (PFS) | Up to 36 months
  PFS is defined as the time from the date of randomization until the first date of documented progressive disease (PD) or death from any cause, whichever occurs first, as measured by RECIST v1.1 using investigator assessments.

SECONDARY OUTCOMES:
Duration of Response (DOR) | Up to 36 months
  DOR is defined as the time from the date of the first documented response until the first date of documented PD or death from any cause, whichever occurs first, as measured by RECIST v1.1 using investigator assessments.
Progression-Free Survival at 6 Months (PFS6) | Up to 6 months
  PFS6 is defined as the proportion of participants alive and PD-free from date of randomization until 6 months as measured by RECIST v1.1 using investigator assessments.
Overall Survival (OS) | Up to 36 months
  OS is defined as the time from the date of randomization until the date of death from any cause.
Overall Survival at 6 Months (OS6) | Up to 6 months
  OS6 is defined as the proportion of participants alive at 6 months from the date of randomization, respectively.
Overall Survival at 12 Months (OS12) | Up to 12 months
  OS12 is defined as the proportion of participants alive at 12 months from the date of randomization, respectively.
Disease Control Rate (DCR) | Up to 36 months
  DCR is defined as the proportion of participants who achieve a CR, PR, or stable disease (SD) as measured by RECIST v1.1 using investigator assessments.
Time to Progression (TTP) | Up to 36 months
  TTP, defined as the time from randomization until the first date of documented PD as measured by RECIST v1.1 using investigator assessments
Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) and Related TEAEs | First dose date up to 24 months plus 100 days
Percentage of Participants Experiencing Clinical Laboratory Abnormalities | First dose date up to 24 months plus 100 days

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (25):
- United States (3):
  - Siteman Cancer Center, St Louis, Missouri
  - Tennessee Oncology, PLLC - Greco-Hainsworth Centers for Research, Nashville, Tennessee
  - The University of Texas, MD Anderson Cancer Center, Houston, Texas
- Australia (4):
  - Monash Health, Clayton, Victoria
  - Alfred Health, Melbourne, Victoria
  - ICON Cancer Center, Kurralta Park
  - Westmead Hospital, Sydney
- China (5):
  - Sichuan Cancer Hospital, Chengdu
  - Zhejiang Cancer Hospital, Hangzhou
  - Guangxi Medical University Cancer Hospital, Nanning
  - Shanghai East Hospital, Shanghai
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
- CHU de Bordeaux, Pessac, France
- Italy (2):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli
- Sarawak General Hospital, Sarawak, Malaysia
- Hospital Universitario Virgen del Rocio, Seville, Spain
- Taiwan (6):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Medical Foundation Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District
- United Kingdom (2):
  - Barts Health NHS Foundation Trust, London
  - The Royal Marsden NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT06727565